CLINICAL TRIAL: NCT03674333
Title: Effect of Adding Folic Acid on Lipid Parameters in Population With Dyslipidemias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Adil Ramzan, Principal Investigator, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1220-5275
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Dyslipidemias
Keywords: Folic Acid; Dyslipidemias; Hyperlipidemia
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: Group A receives Folic Acid and Group B receives Placebo.
Who Masked: Participant
Masking Description: Participants of both the groups will be unaware of whether they received placebo or folic acid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Folic acid 1mg daily will be given to the participants of Group A.
  Interventions: Dietary Supplement: Folic Acid
- Group B (Placebo Comparator): A Placebo (a sugar pill) will be given to the participants of the Group B.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Folic Acid — Folic acid is a water soluble vitamin, required for various biological functions in human body, including metabolism of homocysteine.
  Arms: Group A
Other: Placebo — Placebo - a sugar pill
  Arms: Group B

SUMMARY:
Background: Homocysteinemia is associated with increased risk of stroke, dyslipidemias, dementia, peripheral vascular disease and coronary artery disease. folic acid is involved in the metabolism of homocysteine. Folic acid supplementation helps to reduce homocysteine levels and lowering of homocysteine may cause improvement in serum lipid profile. In this study we will assess the effect of folic acid supplementation for 6 weeks, on lipid parameter in patients who have dyslipidemia.

Methods: It is a placebo controlled randomized trial, consisting of two groups, Group A (n=34) and Group B (n=34). Group A (intervention group) will be given Folic acid supplements and the second group will be given a placebo. After 6 weeks changes in lipid parameters, will be measured in both groups.

Discussion: Folic acid is water soluble vitamin also known as vitamin B-9. Folic acid works as co-factor in many biochemical enzymatic reactions. Homocysteine metabolism also requires folic acid, homocysteinemia may worsen renal function, lipid parameter, accelerate atherosclerosis, angiopathies, and progression of dementia, also increase the risk of stroke and coronary artery disease. In this study, Group A (treatment Group) will be given folic acid supplementation while the Group B (Placebo Group) will be given placebo and at the end of 6 weeks, HDL, LDL, Triglycerides and serum cholesterol levels will be measured and compared with the pre-treatment levels. If Post-treatment group shows significant decrease in serum LDL, total cholesterol, triglycerides and increase in HDL then Folic acid supplementation may be routinely recommended for patient with dyslipidemias.

DETAILED DESCRIPTION:
Hyperlipidemia, increases the risk of stroke, hypertension, coronary artery disease and other associated disorders. World-wide about one-third of coronary artery disease is attributed high cholesterol. Overall it has been estimated that elevated blood cholesterol causes 26 million deaths (4.5% of the total deaths) world-wide. Hyperlipidemias is a major cause of morbidity in both developed and developing countries as a risk factor for stroke and coronary artery disease. The prevalence of raised total cholesterol increased noticeably according to the income level of the country. In low income countries around a quarter of adults had raised total cholesterol, in lower middle income countries this rose to around a third of the population for both sexes. In high-income countries, over 50% of adults had raised total cholesterol; more than double the level of the low-income countries.

Homocysteine, on the other hand, is a sulfur amino acid, which is metabolized by two pathways, either it is re-methylated to methionine or it undergoes trans-sulfuration to cystathionine which is eventually converted into cysteine, an amino acid. Folic acid is involved in remethylation of homocysteine to methionine. Thus, folic acid supplementation may enhance the metabolism of homocysteine level and thereby may decrease its level in blood. Homocysteine in blood is termed as homocysteinemia. Homocysteinemia is associated with dyslipidemias, increased risk of atherosclerosis, micro-angiopathies, coronary artery disease, stroke, dementia and also found to be associated with suppressed immunity. Supplementation with folic acid may lower homocysteine level by accelerating its metabolism to methionine. In this study investigators will be assessing the effect of folate supplementation on the lipid profile, particularly on the blood levels of HDL, LDL, Triglycerides and total cholesterol. The HDL has cardio-protective effect, while on the other hand, the higher level of LDL, total cholesterol and triglycerides may accelerate atherosclerosis, angiopathies and increases the risk of stroke and heart diseases.

Research question: Does addition of folic acid supplementation decrease LDL, total cholesterol, triglycerides and increase HDL in patients with dyslipidemias.

OBJECTIVE:

To assess the effect of folic acid supplementation on HDL, LDL, total cholesterol and triglycerides in patients with dyslipidemias.

HYPOTHESIS Addition of folic acid supplementation will improve lipid parameters (HDL, total cholesterol, triglycerides & LDL) in patients with dyslipidemias.

ELIGIBILITY:
Inclusion Criteria:

* 1. Otherwise, healthy individuals of either sex with any of the following characteristics will be including in the study.

  1. Serum cholesterol >200mg/dl
  2. Serum triglyceride > 150mg/dl
  3. Serum LDL >100mg/dl
  4. Serum HDL < 40mg/dl

Exclusion Criteria:

1. Patients who have any clinically significant or unstable medical or psychiatric illnesses.
2. Patients with CKD, diabetes mellitus, coronary artery disease, with history of stroke, myocardial infarction or any chronic illnesses.
3. Substance abuse such as alcoholism excluded by taking history.
4. Patients who are pregnant are excluded by taking history and urine dipstick test where applicable.
5. Patient who are treated with any investigational drug within last 60 days.
6. Patients who are taking a statin or any other lipid lowering drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-09-24 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
LDL | 6 weeks
  mg/dL
HDL | 6 weeks
  mg/dL
Triglycerides | 6 weeks
  mg/dL
Total Cholesterol | 6 weeks
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Adil Ramzan, MD, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University, Pakistan Institute of Medical Sciences Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data will be available. Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices) will be shared to the researchers who provide a methodologically sound proposal to the primary investigator (Dr. Adil Ramzan).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 5 years following publication of the article.
Access Criteria: Proposal should be directed to "adilramzan@gmail.com". To access data, data requestors will need to sign a data access agreement. Data are available for 5 years at 3rd party website.
URL: http://www.dradilramzan.com

REFERENCES:
- [Background] Blom HJ, Smulders Y. Overview of homocysteine and folate metabolism. With special references to cardiovascular disease and neural tube defects. J Inherit Metab Dis. 2011 Feb;34(1):75-81. doi: 10.1007/s10545-010-9177-4. Epub 2010 Sep 4. PMID 20814827
- [Background] Mierzecki A, Kloda K, Bukowska H, Chelstowski K, Makarewicz-Wujec M, Kozlowska-Wojciechowska M. Association between low-dose folic acid supplementation and blood lipids concentrations in male and female subjects with atherosclerosis risk factors. Med Sci Monit. 2013 Sep 4;19:733-9. doi: 10.12659/MSM.889087. PMID 24002360
- [Background] Baszczuk A, Thielemann A, Musialik K, Kopczynski J, Bielawska L, Dzumak A, Kopczynski Z, Wysocka E. The Impact of Supplementation with Folic Acid on Homocysteine Concentration and Selected Lipoprotein Parameters in Patients with Primary Hypertension. J Nutr Sci Vitaminol (Tokyo). 2017;63(2):96-103. doi: 10.3177/jnsv.63.96. PMID 28552882